CLINICAL TRIAL: NCT01941875
Title: The Effect of Luteal Phase Support on Pregnancy Rate in Intrauterine Insemination Cycles Following Ovarian Stimulation With Gonadotropins
Brief Title: Luteal Phase Progesterone in IUI and Gonadotropin Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032793
Record Dates: First submitted 2013-08-19; First posted 2013-09-13 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Infertility
Keywords: controlled ovarian hyperstimulation; gonadotropins; intrauterine insemination; infertility; luteal progesterone
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Luteal Support (No Intervention): Control group: No luteal phase support or medication will be used
- Luteal Vaginal Progesterone (Experimental): Experiment group: Vaginal progesterone for luteal support beginning the first day after IUI
  Interventions: Drug: Progesterone Effervescent Vaginal Tablets

INTERVENTIONS:
Drug: Progesterone Effervescent Vaginal Tablets — Experimental
  Other Names: Endometrin 100 mg twice daily
  Arms: Luteal Vaginal Progesterone

SUMMARY:
This is a study of patients undergoing Controlled Ovarian Hyperstimulation (COH) with Gonadotropins and Intrauterine Insemination (IUI) at a Fertility Clinic.

Infertility is a common problem, and a popular method of therapy is to inject sperm through the cervix and into the uterus, a procedure known as IUI. In conjunction with IUI, injectable medications (gonadotropins) are used to stimulate the ovaries to produce more than one egg per cycle in a process called COH.

Vaginal progesterone is used for luteal support in in vitro fertilization therapy and has been proven to effect pregnancy rates. However, the role of progesterone in COH is still unclear. In this study, the investigators want to examine the effect of giving vaginal progesterone after COH with IUI on pregnancy rates. The investigators want to study if luteal vaginal progesterone results in a higher pregnancy rate compared to no progesterone therapy in COH with IUI. At present, fertility centres vary in the use of progesterone after insemination, most likely due to the lack of studies on this subject.

At the Fertility Clinic all patients undergoing COH with injectable medications and IUI, regardless of whether they are in the study, have a baseline transvaginal ultrasound and blood tests. Patients start the injectable medications for COH until the ovarian follicles are large enough, then a medication to release the eggs is given. The IUI is done approximately 36 hours later. The day after the IUI, study patients will be given vaginal progesterone while the control patients will receive no progesterone. All patients will be followed until a pregnancy test is done and a viable foetus is confirmed by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Couples with infertility
* Confirmed bilateral tubal patency
* More than 10 million motile sperm available for IUI

Exclusion Criteria:

* Subjects declining enrollment
* Allergies to prescribed vaginal progesterone
* Subjects less than 21 years old or over 43 years old

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | After 6 weeks gestational age
  Presence of a fetal heart beat after 6 weeks gestational age

SECONDARY OUTCOMES:
Biochemical Pregnancy | After 6 weeks gestational age
  Biochemical pregnancy rate
Non-viable Pregnancy | After 6 weeks gestational age
  Non-viable pregnancy rate
Multiple Pregnancy | After 6 weeks gestational age
  Multiple pregnancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility & Womens Endocrine Clinic, Royal Alexandra Hospital, Edmonton, Alberta, Canada